CLINICAL TRIAL: NCT01667185
Title: Effectiveness and Safety of the Dexcom™ G4 Continuous Glucose Monitoring System in Pediatric Subjects With Diabetes Mellitus.
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL900803
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Pediatric Subjects With Diabetes Mellitus
Keywords: pediatric; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric subjects with diabetes mellitus

SUMMARY:
The primary objective of the study is to evaluate the safety and effectiveness of the G4 System (System) when used as an adjuvant to blood glucose testing over a 7-day period in pediatric subjects with diabetes mellitus.

System effectiveness will be primarily evaluated with comparison to laboratory reference Yellow Springs Instrument (YSI) venous sample measurements. The system performance will be evaluated in terms of point and rate accuracy of the system in reference to YSI. The point accuracy is measured as the proportion of G4 System values that are within ±20% of YSI reference value for glucose levels >80 mg/dL and ±20 mg/dL at YSI glucose levels <80 mg/dL. The trend accuracy of the device performance, i.e., continuous glucose error grid analysis, will be evaluated as well as the temporal accuracy at different glucose rates of changes and different glucose ranges (hypoglycemic, euglycemic, and hyperglycemic ranges). The primary matched paired (Sensor-YSI) measurements will be collected during one in-clinic session. System effectiveness will also be evaluated with SMBG measurements similarly.

Safety data of the system will also be collected and safety will be characterized by the incidence of Adverse Device Effects (ADE) experienced by study participants.

Other objectives include the evaluation of device performance at an alternate site (the upper buttocks).

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 17 years ;
* Diagnosis of diabetes mellitus;
* Willing to participate in one 7-day Sensor wear period;
* Willing to wear 2 systems simultaneously;
* Willing to take a minimum of 7 fingersticks per day during home use with a blood glucose meter provided;
* Willing to attend one in-clinic session of up to 6 hours duration. Clinic procedures where blood sampling via SMBG and/or venous YSI method, depending on age;
* Subject or guardian is able to speak, read, and write English.

Exclusion Criteria:

* Extensive skin changes/diseases at sensor wear site that preclude wearing the Sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis);
* Known allergy to medical-grade adhesives;
* Require a magnetic resonance imaging (MRI) scan, computed tomography (CT) scan, or diathermy during the wear period. If any of these procedures are required urgently during the study, subjects will notify the study staff, end their continuous glucose monitoring (CGM) session, and remove their sensor.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
System Performance Effectiveness | 7 days
  The primary objective is to characterize System effectiveness in comparison with the laboratory reference YSI venous sample measurements.

SECONDARY OUTCOMES:
System Performance at Alternate Wear Site | 7 days
  An additional objective is to evaluate System performance at an alternate wear site. The System performance will be assessed, using the same statistical methodology as the primary wear site.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Advanced Metabolic Care and Research, Escondido, California
  - CHOC Children's, Orange, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, Aurora, Colorado
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - Joslin Diabetes Center, Boston, Massachusetts